CLINICAL TRIAL: NCT04900038
Title: A Phase IIb, Randomized, Double-blind, Parallel-group Study to Assess the Efficacy, Safety, Tolerability, and Resistance Profile of GSK3640254 in Combination With Dolutegravir Compared to Dolutegravir Plus Lamivudine in HIV-1 Infected, Treatment-naïve Adults
Brief Title: A Clinical Trial of GSK3640254 + Dolutegravir (DTG) in Human Immunodeficiency Virus-1 Infected Treatment-naive Adults
Acronym: DYNAMIC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company decision to stop compound development. The decision was not based on any safety or efficacy concerns. It reflected the company strategy for portfolio progression.
Sponsor: ViiV Healthcare (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 212483
Record Dates: First submitted 2021-05-19; First posted 2021-05-25 (Actual); Results first posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-11

CONDITIONS: HIV Infections
Keywords: Human immunodeficiency virus-1; GSK3640254; Dolutegravir; Lamivudine; Treatment-naive
MeSH Terms: conditions — HIV Infections | interventions — GSK3640254; dolutegravir; Lamivudine

STUDY DESIGN:
Intervention Model Description: This is a randomized, parallel-group study.
Who Masked: Participant, Investigator
Masking Description: The dose level of GSK3640254 in each of the treatment arms containing GSK3640254 was blinded to the research participants and all study personnel during the study through the Week 24 primary endpoint.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- GSK3640254 100 mg + Dolutegravir (DTG) 50 mg (Experimental): Participants with human immunodeficiency virus type 1 (HIV-1) orally received low dose (100 mg) GSK3640254 tablet blinded and 50 mg DTG unblinded. Each participant received one tablet per day of each intervention up to Week 24.
  Interventions: Drug: GSK3640254; Drug: Dolutegravir
- GSK3640254 150 mg + DTG 50 mg (Experimental): Participants with HIV-1 orally received medium dose (150 mg) GSK3640254 tablet blinded and 50 mg DTG unblinded. Each participant received one tablet per day of each intervention up to Week 24.
  Interventions: Drug: GSK3640254; Drug: Dolutegravir
- GSK3640254 200 mg + DTG 50 mg (Experimental): Participants with HIV-1 orally received high dose (200 mg) GSK3640254 tablet blinded and 50 mg DTG unblinded. Each participant received one tablet per day of each intervention up to Week 24.
  Interventions: Drug: GSK3640254; Drug: Dolutegravir
- DTG 50 mg + Lamivudine (3TC) 300 mg (Active Comparator): Participants with HIV-1 orally received unblinded 50 mg DTG one tablet and blinded 300 mg 3TC. Each participant received one capsule per day of each intervention up to Week 24.
  Interventions: Drug: Dolutegravir; Drug: Lamivudine capsules; Drug: Lamivudine tablets

INTERVENTIONS:
Drug: GSK3640254 — GSK3640254 was available as 25 mg or 100 mg tablets administered orally.
  Arms: GSK3640254 100 mg + Dolutegravir (DTG) 50 mg; GSK3640254 150 mg + DTG 50 mg; GSK3640254 200 mg + DTG 50 mg
Drug: Dolutegravir — DTG was available as 50 mg tablets administered orally.
Drug: Lamivudine capsules — 3TC was available as 300 mg capsules administered orally as a blinded treatment.
  Arms: DTG 50 mg + Lamivudine (3TC) 300 mg
Drug: Lamivudine tablets — 3TC was available as 300 mg tablets administered orally as an unblinded treatment.
  Arms: DTG 50 mg + Lamivudine (3TC) 300 mg

SUMMARY:
The purpose of this study was to evaluate the efficacy of GSK3640254 + DTG relative to lamivudine (3TC) + DTG in treatment-naïve adult participants living with human immunodeficiency virus (HIV)-1. The participants were randomized to one of the three doses of blinded GSK3640254 (100, 150, or 200 milligrams [mgs]) or a reference arm of blinded 3TC-each in combination with open label DTG.

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naive, defined as no anti-retrovirals (ARVs) (in combination or monotherapy) received after a known diagnosis of HIV-1 infection.
* Documented HIV infection and Screening plasma HIV-1 RNA greater than or equal to (>=)1000 c/mL.
* Screening CD4+ T-cell count >=250 cells per millimeter^3 (cells/cubic millimeter).
* Body weight >=50.0 kilograms (kg) (110 pounds [lbs.]) for men and >=45.0 kg (99 lbs.) for women and body mass index (BMI) >18.5 kilograms per meter^2 (kg/meter square). Calculations will utilize sex assigned at birth.

Exclusion Criteria:

* Any evidence of an active Centers for Disease Control and Prevention (CDC) Stage 3 disease [CDC, 2014], except cutaneous Kaposi's sarcoma not requiring systemic therapy.
* Presence of primary HIV infection, evidenced by acute retroviral syndrome (example [e.g.], fever, malaise, fatigue, etc.) and/or evidence of recent (within 3 months) documented viremia without antibody production and/or evidence of recent (within 3 months) documented seroconversion.
* Unstable liver disease (as defined by any of the following: presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice or cirrhosis), known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones or otherwise stable chronic liver disease per investigator assessment);
* History of ongoing or clinically relevant hepatitis within the previous 6 months.
* Any history of significant underlying psychiatric disorder.
* Any history of major depressive disorder with or without suicidal features, or anxiety disorders, that required medical intervention (pharmacologic or not) such as hospitalization or other inpatient treatment and/or chronic (>6 months) outpatient treatment.
* A pre-existing condition, in the opinion of the Investigator or Medical Monitor, that could interfere with normal gastrointestinal anatomy or motility (e.g., gastroesophageal reflux disease [GERD], gastric ulcers, gastritis, inflammatory bowel disease), hepatic and/or renal function, or with the absorption, metabolism, and/or excretion of the study interventions or render the participant unable to take oral study treatment.
* Familial or personal history of long QT syndrome or sudden cardiac death.
* Active treatment for a viral infection other than HIV-1, such as Hepatitis B, with an agent that is active against HIV-1 (were known to be infected with HIV-1 after treatment for Hepatitis B was completed).
* Participants who require concomitant medications known to be associated with a prolonged corrected QT (QTc) interval.
* Exposure to an experimental drug, human blood product, monoclonal antibody, or vaccine (which does not have emergency, conditional, or standard market authorization) within 28 days prior to the first dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2023-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (36):
- United States (8):
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Palm Springs, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Ft. Pierce, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Omaha, Nebraska
- Argentina (2):
  - GSK Investigational Site, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Buenos Aires
- GSK Investigational Site, Montreal, Quebec, Canada
- France (2):
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Tourcoing
- Germany (4):
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Italy (2):
  - GSK Investigational Site, Bergamo, Lombardy
  - GSK Investigational Site, Milan, Lombardy
- Portugal (2):
  - GSK Investigational Site, Porto
  - GSK Investigational Site, Vila Nova de Gaia
- GSK Investigational Site, San Juan, Puerto Rico
- South Africa (4):
  - GSK Investigational Site, Durban
  - GSK Investigational Site, Johannesburg
  - GSK Investigational Site, Parow
  - GSK Investigational Site, Vosloorus Ext 2
- Spain (10):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Bilbao
  - GSK Investigational Site, Elche
  - GSK Investigational Site, La Laguna-Tenerife
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Murcia
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Sant Boi de Llobregat
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Vigo

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Joshi SR, Masia M, Mitha E, Castagna A, Cordova E, Ramgopal M, Gaudion A, Karthika S, Oyee J, Bainbridge V, Wynne B, Lataillade M. Efficacy and safety of the HIV-1 maturation inhibitor GSK3640254 plus dolutegravir as a two-drug regimen in adults naive to antiretroviral therapy (DYNAMIC): 24-week results from a randomised phase 2b study. EClinicalMedicine. 2025 Oct 17;89:103566. doi: 10.1016/j.eclinm.2025.103566. eCollection 2025 Nov. PMID 41357331

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study assessed efficacy, safety and resistance of GSK3640254 in combination with dolutegravir compared to dolutegravir + lamivudine in HIV-1 infected, treatment-naïve adults. The study was terminated by the sponsor after primary analysis (at week 24) as the sponsor determined further development of GSK3640254-containing daily oral regimen would not be differentiated enough from existing 2-drug daily oral regimens. Thus, secondary analyses at week 48 were not evaluated.
Pre-assignment Details: The changes from the planned subsequent analyses were presented as pre-specified in Statistical Analysis Plan. Safety analysis is presented based on the Entire Duration of Treatment Exposure period, which is defined from Day 1 up to end of continued access to treatment post-study termination (Day 478).
Period: Overall Study
Arm/Group | GSK3640254 100 mg + Dolutegravir (DTG) 50 mg | GSK3640254 150 mg + DTG 50 mg | GSK3640254 200 mg + DTG 50 mg | DTG 50 mg + Lamivudine (3TC) 300 mg
Started | 22 | 20 | 22 | 21
Completed | 2 | 3 | 2 | 3
Not Completed | 20 | 17 | 20 | 18
Not completed — Adverse Event | 1 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Study terminated by sponsor | 18 | 15 | 17 | 14
Not completed — Protocol Deviation | 1 | 1 | 0 | 0
Not completed — Participant reached protocol-defined stoping criteria | 0 | 0 | 2 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK3640254 100 mg + Dolutegravir (DTG) 50 mg | GSK3640254 150 mg + DTG 50 mg | GSK3640254 200 mg + DTG 50 mg | DTG 50 mg + Lamivudine (3TC) 300 mg | Total
Number analyzed (Participants) | 22 | 20 | 22 | 21 | 85
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.2 (7.53) | 36.9 (10.51) | 32.6 (8.41) | 32.1 (8.62) | 33.9 (8.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 5 | 3 | 15
  Male | 19 | 16 | 17 | 18 | 70
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 0 | 1 | 1
  Black or African American | 3 | 4 | 3 | 3 | 13
  White | 18 | 14 | 16 | 14 | 62
  Mixed Race | 0 | 1 | 1 | 0 | 2
  Other - Unspecified | 1 | 1 | 2 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Plasma HIV-1 Ribonucleic Acid (RNA) Less Than (<)50 Copies Per Milliliter (c/mL) at Week 24
Description: Percentage of participants with plasma HIV-1 RNA <50 c/mL at Week 24 using the Food and Drug Administration (FDA) snapshot algorithm was assessed to evaluate the antiviral activity in HIV-1 infected ART (anti-retroviral therapy)-naïve participants.
Time Frame: At Week 24
Population: Analysis was performed on Intent-to-Treat Exposed (ITT-E) Population included all randomized participants who received at least one dose of study intervention and had data for plasma HIV-1 RNA <50 c/mL as per timeline assessed.
Measure: Number; unit: Percentage of participants
Groups:
- DTG 50 mg + Lamivudine (3TC) 300 mg: Participants with HIV-1 orally received unblinded 50 mg DTG one tablet and blinded 300 mg 3TC.Each participant received one capsule per day of each intervention up to Week 24.
Arm/Group | GSK3640254 100 mg + Dolutegravir (DTG) 50 mg | GSK3640254 150 mg + DTG 50 mg | GSK3640254 200 mg + DTG 50 mg | DTG 50 mg + Lamivudine (3TC) 300 mg
Number analyzed (Participants) | 22 | 20 | 22 | 21
Percentage of participants | 95 | 85 | 77 | 86

2. Secondary Outcome: Absolute Values of HIV-1 RNA Through Week 24
Description: Plasma samples were collected for quantitative analysis of HIV-1 RNA. Logarithm to base 10 (log 10) values for plasma HIV-1 RNA has been presented. Baseline is defined as the latest non-missing value prior to first dose of treatment according to date and time including unscheduled visits.
Time Frame: At Baseline (Day 1) and Week 24
Population: Analysis was performed on ITT-E Population that had data for absolute values of HIV-1 RNA as per timeline assessed.
Measure: Mean (Standard Deviation); unit: log10 copies per milliliter(log10 c/mL)
Arm/Group | GSK3640254 100 mg + Dolutegravir (DTG) 50 mg | GSK3640254 150 mg + DTG 50 mg | GSK3640254 200 mg + DTG 50 mg | DTG 50 mg + Lamivudine (3TC) 300 mg
Number analyzed (Participants) | 22 | 20 | 22 | 21
log10 copies per milliliter(log10 c/mL)
  Baseline (Day 1) | 4.614 (0.5253) | 4.446 (0.5913) | 4.535 (0.4165) | 4.179 (0.5907)
  Week 24: number analyzed (Participants) | 21 | 19 | 20 | 19
  Week 24 | 1.315 (0.0737) | 1.532 (0.7086) | 1.349 (0.1431) | 1.379 (0.2439)

3. Secondary Outcome: Change From Baseline in HIV-1 RNA Through Week 24
Description: Plasma samples were collected for quantitative analysis of HIV-1 RNA. Logarithm to base 10 (log 10) values for plasma HIV-1 RNA has been presented. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: At Week 24 compared to baseline (Day 1)
Population: Analysis was performed on ITT-E Population that had data for absolute values of HIV-1 RNA as per timeline assessed.
Measure: Mean (Standard Deviation); unit: log10 c/mL
Arm/Group | GSK3640254 100 mg + Dolutegravir (DTG) 50 mg | GSK3640254 150 mg + DTG 50 mg | GSK3640254 200 mg + DTG 50 mg | DTG 50 mg + Lamivudine (3TC) 300 mg
Number analyzed (Participants) | 22 | 20 | 20 | 19
log10 c/mL | -3.306 (0.5163) | -2.874 (0.8476) | -3.186 (0.4809) | -2.767 (0.5531)

4. Secondary Outcome: Absolute Values of Cluster of Differentiation 4+ (CD4+) T-cell Counts Through Week 24
Description: Blood samples were collected and CD4+ cell count assessment by flow cytometry was carried out to evaluate the immunologic activity. Baseline is defined as the latest non-missing value prior to first dose of treatment according to date and time including unscheduled visits.
Time Frame: At Baseline (Day 1) and Week 24
Population: Analysis was performed on ITT-E Population that had data for CD4+ T-cells analysis as per timeline assessed.
Measure: Mean (Standard Deviation); unit: cells per cubic millimeter (cells/mm^3)
Arm/Group | GSK3640254 100 mg + Dolutegravir (DTG) 50 mg | GSK3640254 150 mg + DTG 50 mg | GSK3640254 200 mg + DTG 50 mg | DTG 50 mg + Lamivudine (3TC) 300 mg
Number analyzed (Participants) | 22 | 20 | 22 | 21
cells per cubic millimeter (cells/mm^3)
  Baseline (Day 1) | 436.7 (161.93) | 451.4 (164.86) | 534.8 (200.99) | 506.9 (165.14)
  Week 24: number analyzed (Participants) | 22 | 20 | 19 | 21
  Week 24 | 753.4 (222.73) | 661.0 (193.50) | 756.1 (267.69) | 627.5 (175.94)

5. Secondary Outcome: Change From Baseline in CD4+ T-cell Counts Through Week 24
Description: Blood samples were collected and CD4+ cell count assessment was carried out to evaluate the immunologic activity. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: At Week 24 compared to baseline (Day 1)
Population: Analysis was performed on ITT-E Population that had data for CD4+ T-cells analysis as per timeline assessed.
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | GSK3640254 100 mg + Dolutegravir (DTG) 50 mg | GSK3640254 150 mg + DTG 50 mg | GSK3640254 200 mg + DTG 50 mg | DTG 50 mg + Lamivudine (3TC) 300 mg
Number analyzed (Participants) | 21 | 19 | 19 | 19
cells/mm^3 | 317.7 (175.42) | 200.6 (126.68) | 241.2 (168.83) | 139.5 (126.63)

6. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Deaths, up to End of Continued Access to Treatment Post-study Termination (Day 478)
Description: An SAE is defined as any serious adverse event that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity and is a congenital anomaly/birth defect.
  The study was terminated by the sponsor after primary analysis (at week 24). Adverse event data were collected up to end of continued access to treatment post-study termination (Day 478).
Time Frame: From Day 1 up to end of continued access to treatment post-study termination (Day 478)
Population: Analysis performed on Safety population, that included all randomized participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3640254 100 mg + Dolutegravir (DTG) 50 mg | GSK3640254 150 mg + DTG 50 mg | GSK3640254 200 mg + DTG 50 mg | DTG 50 mg + Lamivudine (3TC) 300 mg
Number analyzed (Participants) | 22 | 20 | 22 | 21
Participants
  SAEs | 2 | 0 | 0 | 1
  Death | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Adverse Events (AEs) Leading to Discontinuation, up to End of Continued Access to Treatment Post-study Termination (Day 478)
Description: Number of participants who discontinued treatment due to AEs are presented. The study was terminated by the sponsor after primary analysis (at week 24). Adverse event data were collected up to end of continued access to treatment post-study termination (Day 478).
Time Frame: From Day 1 up to end of continued access to treatment post-study termination (Day 478)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3640254 100 mg + Dolutegravir (DTG) 50 mg | GSK3640254 150 mg + DTG 50 mg | GSK3640254 200 mg + DTG 50 mg | DTG 50 mg + Lamivudine (3TC) 300 mg
Number analyzed (Participants) | 22 | 20 | 22 | 21
Participants | 1 | 0 | 1 | 0

8. Secondary Outcome: Number of Participants With Adverse Events of Special Interest (AESIs), up to End of Continued Access to Treatment Post-study Termination (Day 478)
Description: AEs of special interest (AESIs) included AEs related to QT prolongation, gastrointestinal (GI) intolerability/toxicity, psychiatric events, nervous system disorders, skin and subcutaneous tissue disorders and cardiac disorders.
  The study was terminated by the sponsor after primary analysis (at week 24). Adverse event data were collected up to end of continued access to treatment post-study termination (Day 478).
Time Frame: From Day 1 up to end of continued access to treatment post-study termination (Day 478)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3640254 100 mg + Dolutegravir (DTG) 50 mg | GSK3640254 150 mg + DTG 50 mg | GSK3640254 200 mg + DTG 50 mg | DTG 50 mg + Lamivudine (3TC) 300 mg
Number analyzed (Participants) | 22 | 20 | 22 | 21
Participants
  AEs related to QT prolongation | 0 | 0 | 0 | 0
  AEs related to GI intolerability/toxicity | 5 | 7 | 8 | 5
  AEs related to psychiatric events | 0 | 3 | 0 | 4
  AEs related to nervous system disorders | 2 | 4 | 5 | 2
  AEs related to skin and subcutaneous tissue disorder | 4 | 0 | 4 | 0
  AEs related to cardiac disorders | 1 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants Who Develop Genotypic Resistance up to Week 24
Description: Blood samples were collected for drug resistance testing to assess the development of viral resistance to GSK3640254 through Week 24. New mutations were tabulated by drug class: integrase strand transfer inhibitor (INSTI), non-nucleoside reverse transcriptase inhibitor (NNRTI), nucleoside reverse transcriptase inhibitor (NRTI) and protease inhibitor (PI).
  Protocol-Defined Virologic Failure (PDVF) was defined as having virologic non-response (HIV-1 RNA <1.0 log10 c/mL reduction from baseline and <200 copies/mL by Week 12, confirmed levels >=200 c/mL at or after Week 24 and plasma HIV-1 RNA <= 50 c/mL from testing on Week 24, virologic rebound (confirmed HIV-1 RNA >=200 copies/mL after confirmed consecutive HIV-1 RNA <50 copies/mL).
Time Frame: From Day 1 up to Week 24
Population: Analysis was performed on ITT-E population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3640254 100 mg + Dolutegravir (DTG) 50 mg | GSK3640254 150 mg + DTG 50 mg | GSK3640254 200 mg + DTG 50 mg | DTG 50 mg + Lamivudine (3TC) 300 mg
Number analyzed (Participants) | 22 | 20 | 22 | 21
Participants | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants Who Develop Phenotypic Resistance up to Week 24
Description: Blood samples were collected for drug resistance testing to assess the development of viral resistance to GSK3640254 and other on-study Anti-Retroviral Therapy (ART) in participants experiencing virologic failure through Week 24. Only plasma HIV-1 RNA values determined by the central laboratory were used to assess virologic failure. PDVF was defined as having virologic non-response (HIV-1 RNA <1.0 log10 c/mL reduction from baseline and <200 copies/mL by Week 12, confirmed levels >=200 c/mL at or after Week 24 and plasma HIV-1 RNA <= 50 c/mL from testing on Week 24, virologic rebound (confirmed HIV-1 RNA >=200 copies/mL after confirmed consecutive HIV-1 RNA <50 copies/mL).
Time Frame: From Day 1 up to Week 24
Population: Analysis was performed on ITT-E Population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3640254 100 mg + Dolutegravir (DTG) 50 mg | GSK3640254 150 mg + DTG 50 mg | GSK3640254 200 mg + DTG 50 mg | DTG 50 mg + Lamivudine (3TC) 300 mg
Number analyzed (Participants) | 22 | 20 | 22 | 21
Participants | 0 | 0 | 0 | 0

11. Secondary Outcome: Trough Concentration (Ctrough) of GSK3640254 at Weeks 2, 4, 8, 12 and 24
Description: Trough concentration (Ctrough) is the concentration reached by a drug immediately before the next dose is administered. This was determined to assess the steady-state exposure of GSK3640254 when given in combination with DTG.
Time Frame: At Weeks 2, 4, 8, 12 (PRE DOSE), 12 (2-6HR POST DOSE), 24 (PRE DOSE), 24 (2-6HR POST DOSE)
Population: Analysis performed on Pharmacokinetic population, which included all participants who received GSK3640254, underwent sparse PK sampling during the study, and provided evaluable GSK3640254 plasma concentration data, demographic and baseline characteristics, and/or information on concomitant medications. Only those participants with data available at specified time points were analyzed for the specific category titles.
Measure: Geometric Mean (95% Confidence Interval); unit: nanogram per milliliter (ng/mL)
Arm/Group | GSK3640254 100 mg + Dolutegravir (DTG) 50 mg | GSK3640254 150 mg + DTG 50 mg | GSK3640254 200 mg + DTG 50 mg
Number analyzed (Participants) | 22 | 20 | 22
nanogram per milliliter (ng/mL)
  Week 2: number analyzed (Participants) | 21 | 19 | 22
  Week 2 | 340.2 [269.5 to 411.0] | 549.9 [390.9 to 708.9] | 724.2 [563.4 to 885.0]
  Week 4: number analyzed (Participants) | 21 | 20 | 21
  Week 4 | 417.8 [330.5 to 505.0] | 632.7 [470.4 to 795.0] | 799.6 [640.9 to 958.3]
  Week 8 | 386.2 [293.7 to 478.6] | 646.6 [421.7 to 871.5] | 821.1 [620.2 to 1022.0]
  Week 12 ( PRE DOSE) | 481.3 [388.6 to 574.0] | 611.4 [430.6 to 792.1] | 877.2 [704.1 to 1050.3]
  Week 12 (2-6HR POST DOSE): number analyzed (Participants) | 21 | 20 | 21
  Week 12 (2-6HR POST DOSE) | 767.8 [612.3 to 923.3] | 1081.2 [759.5 to 1402.8] | 1658.1 [1305.8 to 2010.4]
  Week 24 ( PRE DOSE): number analyzed (Participants) | 21 | 19 | 19
  Week 24 ( PRE DOSE) | 396.0 [331.0 to 460.8] | 570.1 [333.6 to 806.6] | 848.8 [600.3 to 1097.4]
  Week 24 (2-6HR POST DOSE): number analyzed (Participants) | 20 | 20 | 19
  Week 24 (2-6HR POST DOSE) | 759.0 [623.1 to 894.8] | 1107.0 [660.8 to 1553.2] | 1584.1 [1067.3 to 2100.9]

ADVERSE EVENTS:
Time Frame: All cause mortality, non-serious adverse events (Non-SAEs) and serious adverse events (SAEs) were collected up to end of continued access to treatment post-study termination (Day 478).
Description: The study was terminated by the sponsor after primary analysis (at week 24). As prespecified in Statistical analysis plan, AEs were collected up to end of continued access to treatment post-study termination (Day 478).
Arm/Group | GSK3640254 100 mg + Dolutegravir (DTG) 50 mg | GSK3640254 150 mg + DTG 50 mg | GSK3640254 200 mg + DTG 50 mg | DTG 50 mg + Lamivudine (3TC) 300 mg
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/20 | 0/22 | 0/21
Serious Adverse Events (participants affected / at risk) | 2/22 | 0/20 | 0/22 | 1/21
Other Adverse Events (participants affected / at risk) | 16/22 | 15/20 | 17/22 | 14/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3640254 100 mg + Dolutegravir (DTG) 50 mg (N=22) | GSK3640254 150 mg + DTG 50 mg (N=20) | GSK3640254 200 mg + DTG 50 mg (N=22) | DTG 50 mg + Lamivudine (3TC) 300 mg (N=21)
Anogenital dysplasia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3640254 100 mg + Dolutegravir (DTG) 50 mg (N=22) | GSK3640254 150 mg + DTG 50 mg (N=20) | GSK3640254 200 mg + DTG 50 mg (N=22) | DTG 50 mg + Lamivudine (3TC) 300 mg (N=21)
COVID-19 (Infections and infestations) | 3 (3) | 2 (2) | 5 (5) | 3 (3)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastroeneteritis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Monkeypox (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 3 (5) | 3 (3)
Oropharyngeal gonococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pharyngeal chlamydia infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (2) | 2 (2) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory tract infection (Infections and infestations) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 3 (6)
Urethritis chlamydial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 4 (6) | 5 (6) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Faeces soft (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 3 (4) | 3 (3) | 2 (5)
Sciatica (Nervous system disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Blood pressure increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vascular disorders Hypertension (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-08-11): https://cdn.clinicaltrials.gov/large-docs/38/NCT04900038/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-19): https://cdn.clinicaltrials.gov/large-docs/38/NCT04900038/SAP_001.pdf